CLINICAL TRIAL: NCT02175745
Title: 18F-FDOPA PET/CT or PET/MRI in Patients With Gliomas
Brief Title: 18F-FDOPA PET/CT or PET/MRI in Measuring Tumors in Patients With Newly-Diagnosed or Recurrent Gliomas
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Re-evaluate indication with the referring physicians
Sponsor: Erik Mittra (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Erik Mittra, Clinical Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-29364; NCI-2014-01289 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BRN0024 (Other: OnCore); P30CA124435 (NIH)
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Adult Anaplastic Ependymoma; Adult Anaplastic Oligodendroglioma; Adult Brain Stem Glioma; Adult Diffuse Astrocytoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Adult Oligodendroglioma; Adult Pilocytic Astrocytoma; Adult Pineal Gland Astrocytoma; Adult Subependymal Giant Cell Astrocytoma; Childhood High-grade Cerebellar Astrocytoma; Childhood High-grade Cerebral Astrocytoma; Childhood Low-grade Cerebellar Astrocytoma; Childhood Low-grade Cerebral Astrocytoma; Recurrent Adult Brain Tumor; Recurrent Childhood Anaplastic Astrocytoma; Recurrent Childhood Anaplastic Oligoastrocytoma; Recurrent Childhood Anaplastic Oligodendroglioma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Diffuse Astrocytoma; Recurrent Childhood Fibrillary Astrocytoma; Recurrent Childhood Gemistocytic Astrocytoma; Recurrent Childhood Giant Cell Glioblastoma; Recurrent Childhood Glioblastoma; Recurrent Childhood Gliomatosis Cerebri; Recurrent Childhood Gliosarcoma; Recurrent Childhood Oligoastrocytoma; Recurrent Childhood Oligodendroglioma; Recurrent Childhood Pilomyxoid Astrocytoma; Recurrent Childhood Protoplasmic Astrocytoma; Recurrent Childhood Subependymal Giant Cell Astrocytoma; Recurrent Childhood Visual Pathway and Hypothalamic Glioma; Recurrent Childhood Visual Pathway Glioma; Untreated Childhood Anaplastic Astrocytoma; Untreated Childhood Anaplastic Oligoastrocytoma; Untreated Childhood Anaplastic Oligodendroglioma; Untreated Childhood Brain Stem Glioma; Untreated Childhood Cerebellar Astrocytoma; Untreated Childhood Cerebral Astrocytoma; Untreated Childhood Diffuse Astrocytoma; Untreated Childhood Fibrillary Astrocytoma; Untreated Childhood Gemistocytic Astrocytoma; Untreated Childhood Giant Cell Glioblastoma; Untreated Childhood Glioblastoma; Untreated Childhood Gliomatosis Cerebri; Untreated Childhood Gliosarcoma; Untreated Childhood Oligoastrocytoma; Untreated Childhood Oligodendroglioma; Untreated Childhood Pilomyxoid Astrocytoma; Untreated Childhood Protoplasmic Astrocytoma; Untreated Childhood Subependymal Giant Cell Astrocytoma; Untreated Childhood Visual Pathway and Hypothalamic Glioma; Untreated Childhood Visual Pathway Glioma
MeSH Terms: conditions — Ependymoma; Oligodendroglioma; Astrocytoma; Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms; Neoplasms, Neuroepithelial; Optic Nerve Glioma | interventions — fluorodopa F 18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (FDOPA-PET/CT or PET/MRI) (Experimental): Patients receive 18F-fluoro-dihydroxyphenylalanine (18F-FDOPA) intravenously (IV) and then undergo positron emission tomography / computed tomography (PET/CT) or PET/magnetic resonance imaging (PET/MRI) scans 10 to 30 minutes later.
  Interventions: Drug: 18F-fluoro-dihydroxyphenylalanine; Procedure: Positron emission tomography (PET); Procedure: Computed tomography (CT); Procedure: Magnetic resonance imaging

INTERVENTIONS:
Drug: 18F-fluoro-dihydroxyphenylalanine — Administered intravenously (IV)
  Other Names: (18)F-FDOPA; 18F-6-L-fluorodopa; 18F-DOPA; 18F-FDOPA; Fluorine F-18 fluorodopa
Procedure: Positron emission tomography (PET) — Component of an 18F-FDOPA PET/CT or PET/MRI scan
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: Computed tomography (CT) — Component of an 18F-FDOPA PET/CT
  Other Names: tomography, computed; CT scan
Procedure: Magnetic resonance imaging — Component of an 18F-FDOPA PET/MRI
  Other Names: MRI scan; NMR imaging; NMRI; nuclear magnetic resonance imaging

SUMMARY:
To evaluate 18F-FDOPA PET obtained from PET/CT or PET/MRI imaging in patients with newly diagnosed or recurrent gliomas.

DETAILED DESCRIPTION:
This clinical trial compares fluorine F-18 fluoro-dihydroxyphenylalanine (18F-fluorodopa or 18F-FDOPA) positron emission tomography (PET) with standard magnetic resonance imaging (MRI) in measuring tumors in patients with glioma that is newly diagnosed or recurrent (has returned). 18F-FDOPA is a radioactive drug that binds to tumor cells and is captured in images by PET. Computed tomography (CT) and MRI are used with PET to describe information regarding the function, location, and size of the tumor. PET/CT or PET/MRI may be more accurate than standard MRI in helping doctors find and measure brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 15 year-old at the time of radiotracer administration
* Provides written informed consent
* Suspected new diagnosis or suspected recurrence of glioma
* Able to remain still for duration of each imaging procedure (about 20 minutes)

Exclusion Criteria:

* Less than 15 year-old at the time of radiotracer administra
* Unable to provide informed consent
* Inability to lie still for the entire imaging time
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Mittra, MD, PhD, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (FDOPA-PET/CT or PET/MRI): Patients receive 18F-FDOPA intravenously (IV) and then undergo PET/CT or PET/MRI 10-30 minutes later. After completion of study, patients are followed up at 24 hours and at 1 week.
Period: Overall Study
Arm/Group | Diagnostic (FDOPA-PET/CT or PET/MRI)
Started | 2
Completed | 1
Not Completed | 1
Not completed — Not Eligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (FDOPA-PET/CT or PET/MRI)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Suspicious Lesions Identified by 18F FDOPA PET
Description: The number of suspicious lesions will be identified by uptake of F18 FDOPA radiopharmaceutical using a positron emission tomography (PET) scan. Uptake of F-18 FDOPA is a measure of amino acid uptake and metabolism in tumors. Suspicious lesions will be visually identified by a board certified nuclear medicine physician.
Time Frame: Up to 30 minutes after injection of F18 FDOPA
Measure: Number; unit: suspicious lesion(s)
Arm/Group | Diagnostic (FDOPA-PET/CT or PET/MRI)
Number analyzed (Participants) | 1
suspicious lesion(s) | 1

2. Primary Outcome: Percent Agreement of 18F FDOPA PET With Pathology
Description: For the subset of lesions where pathology is available (mainly biopsied lesions), the accuracy of 18F FDOPA PET as percent agreement with pathology will be calculated. If the number of biopsy positive lesions is at least 10, an estimate of sensitivity will be calculate; if the number of biopsy negative lesions is at least 10 an estimate of specificity will be calculated.
Time Frame: Up to 30 minutes post-injection (at time of scan)
Measure: Number; unit: percentage of agreement (sensitivity)
Arm/Group | Diagnostic (FDOPA-PET/CT or PET/MRI)
Number analyzed (Participants) | 1
percentage of agreement (sensitivity) | 100

ADVERSE EVENTS:
Time Frame: 72 Months
Arm/Group | Diagnostic (FDOPA-PET/CT or PET/MRI)
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
This study was underpowered due to low enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No